CLINICAL TRIAL: NCT03711123
Title: A Randomized Controlled Trial of the Effectiveness of Group Metacognitive Therapy vs Clinical Management for Patients With Major Depressive Disorder
Brief Title: Group Metacognitive Therapy vs Clinical Management for Depression
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Oslo (Other)
Responsible Party: Principal Investigator, Toril Dammen, Professor, University of Oslo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015/673-1
Record Dates: First submitted 2018-04-16; First posted 2018-10-18 (Actual); Last update posted 2018-10-18 (Actual); Status verified 2018-10

CONDITIONS: Major Depressive Disorder
Keywords: metacognitive therapy, psychotherapy
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group metacognitive therapy (GMCT) (Experimental): 10 weekly sessions of GMCT With 90 minutes duration
  Interventions: Behavioral: Group metacognitive therapy
- Clinical Management (Active Comparator): 10 weekly individual sessions with up to 60 minutes duration
  Interventions: Behavioral: Clinical management

INTERVENTIONS:
Behavioral: Group metacognitive therapy — 10 weekly Group session of 90 minutes duration
  Arms: Group metacognitive therapy (GMCT)
Behavioral: Clinical management — 10 weekly individual sessions With clinical management including guided self-help
  Arms: Clinical Management

SUMMARY:
The main aims of the study are to (1) compare the effectiveness of Group metacognitive therapy (GMCT) treatment to that of clinical management and (2) explore patterns of change and investigate factors associated with treatment outcome

DETAILED DESCRIPTION:
Major depressive disorder (MDD) is a disabling condition which adversely affects a person's family, work or school life, sleeping and eating habits, and general health.

Cognitive-behavioral therapy (CBT) is a well established effective recommended treatment for MDD. However, only 40-58 % of patients receiving CBT may be classified as recovered using clinical significant change assessed by the Beck Depression Inventory and only between one-third and one quarter of patients receiving CBT remain recovered 18 months after treatment.

A new treatment approach to MDD is Metacognitive Therapy (MCT). In this treatment approach, MDD is conceptualized as being maintained by rumination and meta-cognitions. Treatment seeks to challenge and change specific meta-cognitions and rumination, through behavioural experiments and verbal reattribution. There is accumulating evidence that MCT is effective in the treatment of depression, both individualized and in Groups. A recent pilot study indicated effectiveness above that of CBT. However, the results need to be tested in a randomized controlled trial with a larger sample of patients and a comparison group of active treatment.

The purpose of this trial is to evaluate the effectiveness of Group MCT treatment compared to clinical management included guided self-help and to explore which factors that are associated with depressive symptom outcome in terms of psychological factors, biomarker in terms of heart rate variabilities and polygenic risk score.

The study will be a randomized controlled, trial comprising 64 patients with a primary diagnosis of major depressive disorder (DSM-IV; American Psychiatric Association (APA), 1994). Experienced diagnosticians will assess all patients by using structural interviews such as Structured Clinical Interview for DSM-IV, axis I(SCID I), and axis II disorders (SCID II) and the Hamilton Rating Scale for Depression (HDRS).

All patients will be randomized in blocks to two groups in order to compare the following conditions: Group MCT of 10 weekly sessions lasting 90 minutes and a clinical management condition With 10 weekly individualized sessions up to 60 minutes duration.

Both between-subjects and within-subjects comparisons will be conducted. The research trial will be conducted at an outpatient specialist practice in Drammen, Norway.

The treatment will be administered according to the originators published treatment protocols for MCT for depression. Independent assessors will assess adherence and quality of treatment.

Independent experts will assess the quality of treatment by inspection of a sampling of video-recorded treatments. Using checklists session-by-session will ensure adherence of the therapy. Responsible investigator and supervisors will be using video of all treatment sessions to assess adherence to the treatment condition.

All patients referred for the study will be consecutively assessed at intake (SCID-I + II, HDRS-17). Based on diagnosis and criteria for inclusion and exclusion, the patients will be asked to volunteer to participate in the study and confirm by signing a form of consent.

Patients will be randomized to one of two conditions. Patients will be asked to self-rate symptoms on a battery of self-report questionnaires.

The patients will be assessed prior to treatment, by 10 weeks in treatment, and at six months and at one and two years of follow-up.

Reassessment of the diagnosis and symptom severity is made by post-treatment.

Criteria for recovery will be: Jacobsen criteria of a minimum change and patients crossing the cut-off point on two measures: The HDRS-17 and Beck Depression Inventory (BDI). Other outcome measures will include:

Reduction of depressive symptoms as measured by self-report questionnaires Number of patients with no MDD diagnosis based on SCID-I after treatment Relapse rate during six months and at one and two years follow-up The proportion of responders as measured by the HDRS-17 and BDI and those who no longer fulfil the conditions for a MDD diagnosis after 10 weeks (post-treatment) and by 6 months and one and two years follow-up.

The secondary efficacy variables will be the proportion of responders at 10 weeks (post-treatment) and six months and by one and two years follow-up as measured by the other symptom measures.

A comparison between the two groups of patients will be conducted at 10 weeks (post-treatment) and there will be 6 month and at one- and two years.

A within group analyses will be conducted in order to estimate effect sizes and significant clinical change estimates.

A computer provided by University of Oslo (UiO) will generate the randomization list.

ELIGIBILITY:
Inclusion Criteria:

* MDD is primary problem
* 18-65 years
* stable on medication for at least 8 weeks or medication free
* able to understand and write the Norwegian Language
* signed written informed consent prior to participation

Exclusion Criteria:

* Medical or physical condition underlying depression
* psychosis or organic mental illness
* current suicide intent
* not willing to Accept no changes in medication during treatment
* not willing to Accept random allocation
* cluster A or cluster B personality disorder
* alcohol/substance dependence/abuse
* concurrent psychological treatment or evidence based psychotherapy for depression past year
* bipolar disorder

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2018-11-01 (Estimated); Primary Completion 2021-04 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Change in depression | baseline to 10 weeks (post treatment), 6 months, 12 months and 24 months follow up
  Beck Depression Inventory
Change in diagnosis | baseline to 10 weeks (post treatment), 6 months, 12 months and 24 months follow up
  SCID-I
Change in depression | baseline to 10 weeks (post treatment), 6 months, 12 months and 24 months follow up
  Hamilton Depression Rating Scale 17-item version (HDRS-17) yielding total scores from 0 (least severe) to 52 (most severe)

SECONDARY OUTCOMES:
Change in rumination | baseline to 10 weeks (post treatment), 6 months, 12 months and 24 months follow up
  Ruminative Responses Scale (RRS)
Change in positive beliefs | baseline to 10 weeks, 6 months, 12 months and 24 months follow up
  Positive Beliefs about rumination scale (PBRS)
Change in Negative beliefs | baseline to 10 weeks (post treatment), 6 months, 12 months and 24 months follow up
  Negative beliefs about rumination scale (NBRS)
Change in metacognitions | baseline to 10 weeks (post treatment), 6 months, 12 months and 24 months follow up
  Metacognitions questionnaire-30 (MCQ-30)
Change in personality | baseline to 10 weeks (post treatment), 6 months, 12 months and 24 months follow up
  Distressed type personality (DS-14)
Change in dysfunctional attitudes and beliefs | baseline to 10 weeks (post treatment), 6 months, 12 months and 24 months follow up
  Dysfunctional attitude scales (DAS)
Change in resilience | baseline to 10 weeks (post treatment), 6 months, 12 months and 24 months follow up
  Resilience Scale for adults (RSA)
Change in anxiety | baseline to 10 weeks (post treatment), 6 months, 12 months and 24 months follow up
  Beck Anxiety Inventory (BAI)
Change in sleep | baseline to 10 weeks (post treatment), 6 months, 12 months and 24 months follow up
  Pittsburgh sleep quality inventory (PSQI)
change in report of executive function | baseline to 10 weeks (post treatment), 6 months, 12 months and 24 months follow up
  Behaviour Rating of Executive Function (BRIEF-A)
change in personality diagnoses | baseline to 10 weeks (post treatment), 6 months, 12 months and 24 months follow up
  SCID-II

CONTACTS AND LOCATIONS:
Locations (1):
- Specialist practice Dr Toril Dammen, Drammen, Buskerud, Norway